CLINICAL TRIAL: NCT05037240
Title: Randomized, Placebo-controlled Clinical Trial to Evaluate the Efficacy of an Oral Nutritional Supplement Based on Quercetin in the Prevention of Covid-19 Infection for a Duration of 3 Months
Brief Title: Quercetin in the Prevention of Covid-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1222/01022021
Record Dates: First submitted 2021-09-03; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator)
  Interventions: Dietary Supplement: Quercetin
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin — Quercetin (500 mg), 2 times a day for 3 months
  Arms: Intervention Group
Combination Product: Placebo — 500 mg, 2 times a day for 3 months
  Arms: Placebo

SUMMARY:
Quercetin is a flavonol, a subclass of flavonoid compounds. Of the flavonol molecules, quercetin is the most abundant in fruit and vegetables. Quercetin flavonol is characterized by 3 crucial properties: antioxidant, anti-inflammatory and immunomodulatory. The combination of these 3 properties makes quercetin an excellent candidate for dealing with situations in which oxidative stress, inflammation and the immune system are involved. The purpose of the study is to evaluate the effectiveness of an oral nutritional supplement based on quercetin in the prevention of Covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Absence of Covid-19 infection

Exclusion Criteria:

* Previous Sars-Cov-2 infection demonstrated with antibody positivity through venous sampling
* Demonstrated presence of Sars-Cov-2 through a nasopharyngeal antigenic swab before the start of oral nutritional supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Prevention of Covid-19 infection | Absence of Covid-19 infection at 3 months
  A nasopharyngeal antigenic swab

CONTACTS AND LOCATIONS:
Locations (1):
- Mariangela Rondanelli, Pavia, Italy